CLINICAL TRIAL: NCT03638180
Title: A Double-Blind, Placebo Controlled, Randomized, Adaptive, First-in-Human Study to Assess, Safety, Tolerability, Pharmacokinetics and Food Effect of Single and Multiple Doses of BLU-5937 Administered Orally in Healthy Male and Female
Brief Title: BLU-5937: First-in-Human, Single and Multiple Doses Escalation, Safety, Tolerability, Pharmacokinetics and Food Effect
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bellus Health Inc. - a GSK company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BUS-P5-703
Record Dates: First submitted 2018-08-15; First posted 2018-08-20 (Actual); Last update posted 2018-11-09 (Actual); Status verified 2018-08

CONDITIONS: Cough
MeSH Terms: conditions — Cough | interventions — BLU-5937

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Single Ascending Doses (Experimental): Single ascending doses, 6 dose levels
  Interventions: Drug: BLU-5937; Drug: Placebo
- Multiple Ascending Doses (Experimental): Multiple ascending doses, 3 dose levels
  Interventions: Drug: BLU-5937; Drug: Placebo

INTERVENTIONS:
Drug: BLU-5937 — BLU-5937 oral tablet
Drug: Placebo — Matching placebo to BLU-5937

SUMMARY:
This is a first-in-human study that will investigate the safety, tolerability and pharmacokinetics of ascending single and multiple doses of BLU-5937 using a double blind, placebo controlled, randomized, adaptive, single center study design. The influence of food on the pharmacokinetics of BLU-5037 will also be investigated.

DETAILED DESCRIPTION:
BLU-5937 is a selective P2X3 receptor antagonist being developed for the treatment of chronic cough. This Phase 1 study will investigate the safety, tolerability and pharmacokinetics of ascending single and multiple doses of BLU-5937 administered orally to healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult male and/or female (non-childbearing potential or, for women of childbearing potential, using 2 forms of acceptable birth control or agreed to abide by true abstinence),
* Age: 18 to 55 years (inclusive).
* Body mass index (BMI) : ≥18.5 and ≤30 kg/m².
* Non or ex smoker.

Exclusion Criteria:

* Any findings from the medical examination (including medical history, physical examination, vital signs, laboratory tests and ECG) outside from normal and deemed by the investigator to be clinically significant.
* Use of any prescription drugs (with the exception of hormone replacement therapy) in the 28 days prior to the first study drug administration, that in the opinion of the investigator would put into question the status of the volunteer as healthy.
* Volunteers who took an Investigational Product in the 28 days prior to the first study drug administration.
* Volunteers who donated 50 mL or more of blood in the 28 days prior to the first study drug administration.
* Donation of 500 mL or more of blood in the 56 days prior to the first study drug administration.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2018-07-09 (Actual); Primary Completion 2018-10-25 (Actual); Study Completion 2018-10-25 (Actual)

PRIMARY OUTCOMES:
Number and severity of treatment emergent adverse events (TEAEs) | up to 48 hours after the last dose
  Number and severity of TEAEs collected from dosing until follow up 48 hours after last dose

SECONDARY OUTCOMES:
Maximum plasma concentration (Cmax) | up to 48 hours after the last dose
  To assess Cmax of single and multiple ascending oral doses of BLU-5937
Area under the curve (AUC) | up to 48 hours after the last dose
  To assess AUC of single and multiple ascending oral doses of BLU-5937
Maximum plasma concentration (Cmax) under fed conditions | up to 48 hours after the last dose
  To assess Cmax of a single oral dose of BLU-5937 under fed conditions
Area under the curve (AUC) under fed conditions | up to 48 hours after the last dose
  To assess AUC of a single oral dose of BLU-5937 under fed conditions

CONTACTS AND LOCATIONS:
Locations (1):
- Alta Sciences Algorithme Pharma, Mount Royal, Quebec, Canada